CLINICAL TRIAL: NCT01953042
Title: A Randomized Trial Testing the Benefits of a Psychoeducation Program for Those Awaiting Treatment for OCD and OCD Spectrum Disorders
Brief Title: Benefits of a Psychoeducation Program for Those Awaiting Treatment for OCD and OCD Spectrum Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of dedicated resources at this time.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Neil Rector, Research Scientist, Psychologist, and Director of the Mood and Anxiety Treatment and Research Program, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 279-2013
Record Dates: First submitted 2013-09-25; First posted 2013-09-30 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Obsessive-Compulsive Disorder; Anxiety Disorders
Keywords: Obsessive-Compulsive Disorder; Health Education
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waitlist as Per Usual (No Intervention): Wait list as per usual with no additional information sessions
- Waitlist and Psychoeducation (Active Comparator): Patients remain on waitlist but also receive 4 additional educational sessions (8 hours each)
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — 4 educational sessions covering information on diagnosis, treatment, available resources and self care for OCD and OCD Spectrum Disorders
  Arms: Waitlist and Psychoeducation

SUMMARY:
This study will examine the effect of offering information sessions to a randomized group of patients with OCD spectrum disorders. Psychoeducation is a component of first line treatment; though intended to be informative in nature, these psychoeducation services can have a positive effect on quality of life, sense of self-efficacy, functioning and a person's readiness to engage in long term treatment. However, no studies have dismantled and tested the independent effect of psychoeducation from standard treatment such as Cognitive Behavioural Therapy. This study aims to directly test the potential effect of one aspect of CBT that if found to be helpful, can become a distinct early intervention component of care so that as people await services, they can profit from the early benefits associated with attending these information sessions. This study therefore sets out to examine the potential early benefits of providing education about the illness on symptom functioning, quality of life and readiness to engage in more formal treatment. We will offer 4 structured information sessions to individuals allocated to a wait list for services related to the treatment of OCD and OCD Spectrum Disorders in order to directly test the benefit of adding a didactic structured psychoeducation program to our services. The study will be a randomized trial where subjects (N=50) will be randomly assigned to receive either 1) 4 educational sessions covering information on diagnosis, treatment, available resources and self care for OCD and OCD Spectrum Disorders or 2) wait list as per usual with no additional information sessions. The experimental design is a 2 (treatment condition) by 2 (assessment phase) repeated measures factorial design. It is hypothesized that subjects participating in the psychoeducation group compared to the wait list control group will see greater reductions in self-reported measures of symptom severity and improvement in other measures of quality of life, level of functioning, self-efficacy and readiness to engage in treatment. If this study can demonstrate that the addition of a short structured informative intervention of 4 sessions can confer early benefits for those suffering with OCD and OCD spectrum disorders, then it provides another route by which patients can improve this condition specifically while waiting for consultation and the opportunity to receive a more structured, evidence-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Referred for treatment services at the Frederick W. Thompson Anxiety Disorder Centre at Sunnybrook Health Sciences Centre
* Presenting with OCD or OCD Spectrum Disorders
* Ability to communicate in written and spoken English

Exclusion Criteria:

* Active substance abuse/dependence
* Suspected organic pathology
* Recent suicide attempt/active suicideality
* Active bipolar or psychotic disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity from Baseline in OCD and Spectrum Measures | 4 months
  OCD measures will include the 18-item Obsessive Compulsive Inventory-Revised (OCI-R), measuring subscales of Washing, Checking, Doubting, Ordering, Obsessions, Hoarding and Neutralizing, as well as a self-report version of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS-SR), a 3 part questionnaire containing a 58 item symptom checklist, identification of the most prominent obsessions and compulsions and a 10 item severity scale. OCD Spectrum measures will include the Body Dysmorphic Disorder-YBOCS, Savings Inventory Revised, PITS, and the MGH scale.

SECONDARY OUTCOMES:
Change in Quality of Life from Baseline | 4 months
  Measures capturing quality of life, level of impairment, self-efficacy, and readiness to change will include the Quality of Life Enjoyment Questionnaire (Q-LES-Q-SF), the Sheehan Disability Scale, the Illness Intrusiveness Rating Scale (III), the University of Rhode Island Change Assessment (URICA), the SF-36, and the COPE Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Rector, Ph.D., C.Psych., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No